CLINICAL TRIAL: NCT05102604
Title: A Pilot Study to Determine the Effect of Avocado Consumption on Skin Aging
Brief Title: The Effect of Avocado vs. Usual Diet on Skin Aging
Acronym: AvoSkin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Hass Avocado Board (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-001834
Record Dates: First submitted 2021-08-24; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Skin Inflammation
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two equally sized groups.
Masking Description: Both groups will be instructed to continue to follow their habitual diet but the intervention group will receive one avocado per day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avocado (Active Comparator): one avocado per day
  Interventions: Other: Avocado
- Habitual Diet (Placebo Comparator): maintain habitual diet
  Interventions: Other: Habitual diet

INTERVENTIONS:
Other: Avocado — Subjects will eat one avocado in addition to their usual diet
  Arms: Avocado
Other: Habitual diet — Subjects will eat their usual diet
  Arms: Habitual Diet

SUMMARY:
This clinical trial aims to assess the effect of providing one avocado per day on skin health in comparison with a control group maintaining their habitual diets. Participants will be randomly assigned to one of two equally sized groups. Both groups will be instructed to continue to follow their habitual diet but the intervention group will receive one avocado per day. Participants will be followed for outcomes for a four-month period.

DETAILED DESCRIPTION:
This study will be a randomized, parallel group comparison of daily avocado consumption vs. habitual diet. The study will be carried out in accordance with the guidelines of the Human Subjects Protection Committee of the University of California, Los Angeles. All subjects will give written informed consent before the study begins.

At screening, informed consent and HIPAA authorization will be reviewed and signed. A medical history will be obtained. Enrollment will be reviewed by the study physician according to inclusion and exclusion criteria. Skin type and response to UVB will be assessed.

At baseline, participants will undergo skin testing. Subjects will consume 1 avocado a day (Hass Avocado) or maintain habitual diet (up to 2 avocados/month) daily for 16 weeks. Skin will be assessed at weeks 0, 8 and 16. Each group will have 20 subjects as calculated by power analysis. Two additional subjects for each group will be recruited for possible dropouts and a total of 22 subjects will be recruited for each group.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects
* Increased waist circumference defined as ≥35 inches for women (NCEP ATP III 2005)
* Women
* At least 25 years old at screening
* Not currently eating more than 2 avocados per month (habitual intake in U.S.)
* Non-smokers
* Fitzpatrick Skin type II-IV
* Willing to maintain their normal skin care pattern for the duration of the study (avoiding excessive sun, not beginning new skin treatments)
* Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment

Exclusion Criteria:

* Does not eat avocados
* Sensitive / allergic to avocados
* Allergies to latex or oral allergy syndrome
* Not willing or unable to undergo MRI scans
* Unstable medical condition such as on dialysis for renal disease, cardiac, gastrointestinal, or hepatic disease, cancer (non-melanoma skin cancer >5 years ago acceptable, any cancer site >10yrs without recurrence).
* Pregnant, lactating, intention of pregnancy
* Lost or gained 10 lbs of body weight in last year
* Following restricted or weight loss dietary patterns
* Subjects who cannot avoid excessive exposure to either natural or artificial sunlight.
* Unstable anti-anxiety / anti-depressive / anti-psychotic medication use defined as dose change within last 6 months
* Currently taking any prescription medications that increase the risk of photosensitivity or history of taking such medications in the less than 3 months (e.g. alpha-hydroxy acids in cosmetics, antibiotics (ciprofloxacin, doxycycline, levofloxacin, ofloxacin, tetracycline, trimethoprim), antifungals (flucytosine, griseofulvin, voricanozole), antihistamines (cetirizine, diphenhydramine, loratadine, promethazine, cyproheptadine), Accutane
* Oral steroid use within the last 6 months longer than 7 days
* Elevated alcohol intake (7+ drinks/week females; 14+ drinks/week males)
* Participation in another clinical intervention trial within 30 days of baseline

Ages: 25 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Minimal erythema | 16 weeks
  Standardized inflammation will be induced by irradiating test areas on the inner arm of subjects with defined doses of narrow band ultraviolet B (NB-UVB) light delivered by the Dermalight 90 handheld device (National Biological).
Skin Elasticity | 16 weeks
  The Cutometer measures the vertical deformation of the skin in millimeters when the skin is pulled by means of a controlled vacuum into the circular aperture, 6mm in diameter, of the probe. In its standard configuration, the Cutometer is equipped with a measuring probe with a 2mm aperture because the device is originally designed to measure only the elastic properties of the epidermis. Skin hydration will measured using the moisture/hydration probe that attaches to the Cutometer. We will measure six sites: forehead, under the eye, frontal cheek, crow's foot, lateral cheek, and inner forearm.

SECONDARY OUTCOMES:
Skin Type Classification | 16 weeks
  Developed in 1975, the system classifies skin type according to the amount of pigment the skin has and the skin's reaction to sun exposure. This information can help predict your overall risk of sun damage and skin cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No